CLINICAL TRIAL: NCT05214521
Title: Investigation of the Effectiveness and Safety of Rehabilitation of Patients With Impaired Fine Function of the Hand Due to a Stroke Using "Glove Simulator "SensoRehab" Based on Digital Interactive Technologies With Artificial Intelligence
Brief Title: Digital Interactive Technologies in Rehabilitation of Post-sroke Patients With Impaired Fine Function of the Hand
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Moscow Scientific and Practical Center of Medical Rehabilitation, Restorative and Sports Medicine (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 9 12112020
Record Dates: First submitted 2022-01-14; First posted 2022-01-28 (Actual); Last update posted 2022-05-17 (Actual); Status verified 2022-05

CONDITIONS: Stroke Rehabilitation
Keywords: post-stroke dysfunction of the hand; upper limb medical rehabilitation; digital interactive technology; artificial intelligence; ischemic stroke rehabilitation

STUDY DESIGN:
Intervention Model Description: an open-label observational trial
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- digital interactive technology Smart glove "SensoRehab" (Experimental): The operation of the digital interactive complex Smart glove "SensoRehab" is based on the visual and kinesthetic (proprioceptive) biofeedback principle by using a set of cognitive interactive computer games controlled by finger and hand movements. The technique involves neurosensory training and retraining to improve the fine use of the hand and arm, and the patient's cognitive and emotional state.
  Interventions: Device: digital interactive technology Smart glove "SensoRehab"

INTERVENTIONS:
Device: digital interactive technology Smart glove "SensoRehab" — Participants will receive rehabilitation program including sessions on the Smart glove "SensoRehab" (SGSR) system. The program for IS patients includes 10 sessions with the SGSR: 15-30 minutes once a day for the affected hand, 2 weeks.

SUMMARY:
The aim of the study is to investigate the efficacy and safety of digital interactive technology with artificial intelligence and biofeedback Smart glove "SensoRehab" for restoration of in-hand manipulation in patients with ischemic stroke in the early and late recovery periods.

DETAILED DESCRIPTION:
The study is an open-label observational trial. Brain stroke (BS) is one of the main causes of upper limb (UL) dysfunction and limitations of daily human activity.The fine use of the hand imparement is often combined with speech, cognitive and emotional disturbances, which is due to the anatomical proximity and close functional relationships of the corresponding areas in the cerebral cortex.

The objective of the present study will be to evaluate the effectiveness and safety of the digital interactive technology (DIT) with artificial intelligence and biofeedback Smart glove "SensoRehab" (SGSR) for restoration of in-hand manipulation in patients with ischemic stroke in the early and late recovery period.The SGSR technique involves neurosensory training and retraining to improve the fine use of the hand and arm, and the patient's cognitive and emotional state.

30 patients will be include to the study. After a basic assessment of hand motor function and game training, each patient undergoes sessions on the SGSR system. The program for BS patients includes 10 sessions with the SGSR (15-30 minutes once a day for the affected hand, 2 weeks).

The clinical outcomes will be obtained at the completion of treatment (2 weeks) and at 1 month after ompletion of the course of rehabilitation. The statistical analysis will follow the intention-to-treat principles.

The outcomes of interest are motor function state of the UL, pain intensity, cognitive functions, general physical and emotional status. An integral indicators are the assessment of the patient's quality of life and independence in everyday life activity.

ELIGIBILITY:
Inclusion Criteria:

1. Men or women aged 18 to 70 years after a first-onset IS, early (1-6 months), late recovery (6-12 months) periods.
2. Supratentorial IS according to MRI of the brain.
3. The severity of UL paresis ranged from a score of 4 to 3 according to the Medical Research Council Scale (MRCS).20
4. Spasticity of 2 points or less by the Modified Ashworth Scale (MAS)
5. Cognitive function more than 20 points on the Montreal Cognitive Assessment (MoCA)
6. Affective disorders score less than 11 on the Hospital Anxiety and Depression Scale (HADS)
7. The patient's ability and willingness to comply with the requirements of this protocol.

Exclusion Criteria:

1. Concomitant neurological diseases causing decreased muscle strength or increased muscle tone in the UL (e.g., cerebral palsy, brain injury).
2. Clinically significant limitation of the passive movement amplitude in the joints of the investigated hand, pronounced contracture and deformities of the upper extremity.
3. Use of other DIT, BFB techniques to restore impaired UL function within 30 days prior to the patient Inclusion Visit.
4. Severe visual impairment, decreased visual acuity of less than 0.2 in the worst eye according to the Golovin-Sivtsev Table24.
5. Sensory aphasia, gross motor aphasia.
6. Recurrent stroke.
7. Unstable angina and/or heart attack in previous month.
8. Uncontrolled arterial hypertension.
9. Somatic diseases in decompensation stage.
10. Alcohol abuse, medical marijuana use or soft drug abuse within the 12 months prior to the Inclusion Visit.
11. Any medical condition, including mental disease or epilepsy that could affect the interpretation of study results, the study procedures or patient safety.
12. Pregnancy.
13. Lactation.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2021-01-11 (Actual); Primary Completion 2022-12-30 (Estimated); Study Completion 2023-12-30 (Estimated)

PRIMARY OUTCOMES:
Fugl-Meyer Upper Extremity Scale (FMA-UE) dynamic | Baseline, end of the 2-nd week
  The FMA UE Scale comprises 33 items, each scored on a scale of0 to 2, where 0 = cannot perform, 1 = performs partially and2 = performs fully. It is free, requires only household items fortesting, and takes up to 30 minutes to administer. Changes in sections A-D of the FMA-UE Scale by 7 points or more are considered as efficacy.
Fugl-Meyer Upper Extremity Scale (FMA-UE) dynamic | Baseline, 1-month after completing training
  The FMA UE Scale comprises 33 items, each scored on a scale of0 to 2, where 0 = cannot perform, 1 = performs partially and2 = performs fully. It is free, requires only household items fortesting, and takes up to 30 minutes to administer. Changes in sections A-D of the FMA-UE Scale by 7 points or more are considered as efficacy.
Action Research Arm Test (ARAT) Scale dynamic | Baseline, end of the 2-nd week
  The Action Research Arm Test (ARAT) is a 19 item observational measures. Items comprising the ARAT are categorized into four subscales (grasp, grip, pinch and gross movement) and arranged in order of decreasing difficulty, with the most difficult task examined first, followed by the least difficult task. Task performance is rated on a 4-point scale, ranging from 0 (no movement) to 3 (movement performed normally). Changes in the total ARAT Scale score by 4 points or more more are considered as efficacy.
Action Research Arm Test (ARAT) Scale dynamic | Baseline, 1-month after completing training
  The Action Research Arm Test (ARAT) is a 19 item observational measures. Items comprising the ARAT are categorized into four subscales (grasp, grip, pinch and gross movement) and arranged in order of decreasing difficulty, with the most difficult task examined first, followed by the least difficult task. Task performance is rated on a 4-point scale, ranging from 0 (no movement) to 3 (movement performed normally). Changes in the total ARAT Scale score by 4 points or more more are considered as efficacy.

SECONDARY OUTCOMES:
percentage of correctly performed tasks | Baseline, end of the 2-nd week
  percentage of correctly performed tasks while training
change in the paresis degree The 6-point Medical Research Council Scale for assessing muscle strength: MRCS | Baseline, end of the 2-nd week and 1-month after completing training
  The 6-point Medical Research Council Scale for assessing
changes in spasticity severity | Baseline, end of the 2-nd week and 1-month after completing training
  Modified Ashworth Scale: MAS (0 to 4 points)
changes in level of impairment or dependence in daily life | Baseline, end of the 2-nd week and 1-month after completing training
  Barthel ADL Index
сhanges in cognitive status | Baseline, end of the 2-nd week and 1-month after completing training
  Montreal Cognitive Assessment: МоСА
Presence and severity of depression | Baseline, end of the 2-nd week and 1-month after completing training
  The Hospital Anxiety and Depression Scale: HADS. Changes in HADS anxiety and depression scores
Life quality assessment | Baseline, end of the 2-nd week and 1-month after completing training
  European Quality of Life Questionnaire EuroQol EQ-5D-5L (version 1.0, 2011 in combination with the visual analogue scale)

CONTACTS AND LOCATIONS:
Overall Officials: Elena V Kostenko, MD, Principal Investigator — Moscow Scientific and Practical Center of Medical Rehabilitation, Restorative and Sports Medicine
Locations (1):
- Moscow Scientific and Practical Center of Medical Rehabilitation, Restorative and Sports Medicine, branch 7, Moscow, Russia